CLINICAL TRIAL: NCT05948007
Title: The Role of Neurofeedback Training and Pain Management in Post-operative Shoulder Rehabilitation: a Study Connecting Neural Mechanism and Clinical Results
Brief Title: The Role of Neurofeedback Training and Pain Management in Post-operative Shoulder Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Poyu Chen, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202102407B0
Record Dates: First submitted 2023-06-04; First posted 2023-07-17 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Pain, Shoulder; Post Operative Pain
Keywords: Shoulder pain; Post operative pain; Pain management; Neurofeedback
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: All participants will receive any medical care they would normally receive, including post-surgery exercise program. Those randomized to the usual care group are free to seek whatever treatment, if any, they would like to take.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neurofeedback group (Experimental): 12 training sessions within 6 weeks, starting with FAA modulation followed by the frontal midline theta upregulations.
  Interventions: Device: Neurofeedback training
- Sham neurofeedback group (Sham Comparator): Same dosage as the neurofeedback group
  Interventions: Device: Sham-neurofeedback training
- Pain management protocol (Active Comparator): The PMP includes cognitive behavioral therapy techniques, and pain neuroscience education.
  Interventions: Behavioral: Pain management protocol
- Care as usual (No Intervention): Providing medical care as they would normally receive, including a post-surgery exercise program.

INTERVENTIONS:
Device: Neurofeedback training — 12 training sessions within 6 weeks will be provided. In each training session, participants will have neurofeedback training for five 3-minute training periods.
  Arms: Neurofeedback group
Device: Sham-neurofeedback training — The Sham group has the same training dosage as the neurofeedback group.
  Arms: Sham neurofeedback group
Behavioral: Pain management protocol — The treatment components include sleep psychoeducation, sleep hygiene education, exercise consultation, and cognitive-behavioral pain management, i.e., practice in changing dysfunctional thoughts, setting and working toward behavioral goals, relaxation skills
  Arms: Pain management protocol

SUMMARY:
The primary aim is to compare the efficacy of neurofeedback training (NFT) and pain management protocol (PMP) in pain reduction, restoration of shoulder function, and improved cognitive performance as the post-operative rehabilitation protocols in shoulder pain patients.

DETAILED DESCRIPTION:
The primary aim is to compare the efficacy of neurofeedback training (NFT) and pain management protocol (PMP) in pain reduction, restoration of shoulder function, and improved cognitive performance as the post-operative rehabilitation protocols in shoulder pain patients. While the former modulates neural activity, the latter focuses on biopsychosocial aspects of pain, respectively. Also, we will measure the peripheral cytokine levels of rotator cuff injury to clarify the possible role of peripheral inflammation on central neural activities. By incorporating the behavior (both motor and cognition), peripheral inflammation, and neural activity, we believe this study would bridge the gap between mind and body as the "whole person" approach to understanding musculoskeletal pain and its appropriate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pain ≥3months and ≥3 days per week
* Pain intensity ≥ 40 (VAS scale from 0 no pain to 100 very painful)
* Participants in the neurofeedback training group and pain management group were asked not to involve other treatment when they are in the 6th-12th week intervention period.
* The surgical indication would be based on orthopedics opinions.

Exclusion Criteria:

* shoulder surgery in the prior 3 years
* osteoporotic vertebral fractures or rheumatologic diseases
* chronic wide- spread pain syndromes (fibromyalgia or chronic fatigue syndrome)
* pain at any other location in addition to shoulder pain
* Neurological disease, i.e., stroke, parkinson's disease, etc..
* Cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Pain-related measurement 1: Changes of Visual Analogue Scale (VAS) | pre-operative (T0), before and after each training session over 6 week period, and post-operative 12 weeks (T1)[As after training], and post-operative 24 weeks (T2) [As follow-up]
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Neuropsychological assessment 1: Changes of Montreal Cognitive Assessment (MoCA) | pre-operative (T0), and post-operative 24 weeks (T2) [As follow-up]
  The MoCA assesses general cognitive ability. Scores range from 0 to 30. Higher scores denote better cognitive function.
Neurophysiology recording 1: Changes of resting EEG oscillatory | pre-operative (T0), and post-operative 24 weeks (T2) [As follow-up]
  Brain activity will be recorded continuously

SECONDARY OUTCOMES:
Disease-specific outcome measurement 1: Changes of American Shoulder and Elbow Surgeons Assessment (ASES) | pre-operative (T0), post-operative 12 weeks (T1) [As after training], and post-operative 24 weeks (T2) [As follow-up]
  The ASES is a reliable and validated questionnaire that evaluates functional limitations in patients with shoulder dysfunction. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Disease-specific outcome measurement 2: Changes of Constant Score (CS) | pre-operative (T0), post-operative 12 weeks (T1) [As after training], and post-operative 24 weeks (T2) [As follow-up]
  The CS is a reliable and valid measurement specifically designed for evaluating shoulder joint function. The maximum possible score on the CS is 100, with higher scores indicating better overall shoulder function.
Disease-specific outcome measurement 3: Changes of the health state of EQ-5D-5L | pre-operative (T0), post-operative 12 weeks (T1) [As after training], and post-operative 24 weeks (T2) [As follow-up]
  The questionnaire of EQ-5D-5L comprises 5 dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores of each dimension range from 1 (no problem) to 5 (unable to/extreme problems); whereas, the numerical description of 5-dimension questionnaire represents the health state.
Mood-related measurement 1: Changes of Beck Depression Inventory II (BDI-II) | pre-operative (T0), post-operative 12 weeks (T1) [As after training], and post-operative 24 weeks (T2) [As follow-up]
  The BDI-II is a well-validated questionnaire that assesses the severity of depressive symptoms. The total score ranges from 0 to 63, with higher scores indicating more severe depressive symptoms.
Mood-related measurement 2: Changes of State-Trait Anxiety Inventory (STAI) | pre-operative (T0), post-operative 12 weeks (T1) [As after training], and post-operative 24 weeks (T2) [As follow-up]
  The STAI is a widely used measure of anxiety that consists of two scales: the STAI-S measures state anxiety, which assesses the individual's current emotional condition, and the STAI-T measures trait anxiety, which reflects the person's stable tendency to experience anxiety. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Subjective sleep quality 1: Changes of Pittsburgh Sleep Quality Index (PSQI) | pre-operative (T0), post-operative 12 weeks (T1) [As after training], and post-operative 24 weeks (T2) [As follow-up]
  The PSQI is a widely used and reliable questionnaire that evaluates sleep quality over the past month. Scores range from 0 to 21, with lower scores indicating healthier sleep quality.
Objective sleep quality | pre-operative (T0), post-operative 12 weeks (T1) [As after training], and post-operative 24 weeks (T2) [As follow-up]
  Actigraphy with an ambient light sensor
Neuropsychological assessment 2: Changes of subjective cognitive declince | pre-operative (T0), and post-operative 24 weeks (T2) [As follow-up]
  Everyday Cognition (Ecog-12) assesses general subjective cognitive decline. Scores range from 12 to 24. The score of 14 or above indicates subjective cognitive decline.
Neuropsychological assessment 3: Changes of Digit Symbol Coding from Wechsler Adult Intelligence Scale III (WAIS-III) | pre-operative (T0), and post-operative 24 weeks (T2) [As follow-up]
  Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time (e.g. 90 or 120 sec) is measured. The more the number of correct symbols, the better the speed of processing.
Neuropsychological assessment 4: Changes of Digit Span from Wechsler Adult Intelligence Scale IV (WAIS-IV) | pre-operative (T0), and post-operative 24 weeks (T2) [As follow-up]
  The test consists of three parts: forward span, backward span, and sequencing. In the forward span, the participant is asked to repeat the numbers read in one second intervals following the same order; whereas, in the backward span, the participant is requested to repeat the numbers read in one second intervals in reverse order from the end to the beginning. In the sequencing, the participant is asked to recall and repeat the numbers read in one second intervals in ascending order. The highest score that can be obtained for each part is 16 points, with a total score of 48 points. A higher point indicates better working memory.
Neuropsychological assessment 5: Changes of the times in Color Trials Test (CTT) | pre-operative (T0), and post-operative 24 weeks (T2) [As follow-up]
  The CTT is a cognitive assessment tool by connecting numbered circles and color in sequence. The test consists of two parts: CTT 1 (connecting numbered circles from 1 to 25) and CTT 2 (connecting numbered circles from 1 to 25 alternating between two colors). The times in CTT 1 and CTT 2 will be measured respectively. The lesser time indicates greater cognitive flexibility and processing speed.

OTHER OUTCOMES:
Pain-related measurement 3: Tampa Scale of Kinesiophobia (TSK-11) | pre-operative (T0)
  The TSK is one of the most frequently employed measures for assessing pain-related fear in patients with chronic musculoskeletal pain. The 11-item TSK total scores range from 11 to 44 where the lowest 11 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Pain-related measurement 4: Pain Catastrophizing Scale (PCS) | pre-operative (T0)
  The PCS is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with pain or not.
Cytokine from Joint fluid (JF) | at the beginning of the surgery
  The aspiration procedures will be performed immediately prior to the creation of skin incisions in the operating room by surgeons under anesthesia. The samples will be transferred to sealed vials, then frozen and stored at 80°C until analysis. The JF samples (50, 100 and 200 lL) will be subjected to measurements of IL-1b, IL-6 and IL-8 levels using ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Poyu Chen, PhD, Study Chair — Chang Gung University